CLINICAL TRIAL: NCT01673451
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of E2006 in Healthy Adult and Elderly Subjects
Brief Title: 2-Part Multiple Ascending Dose Study for Safety and Pharmacokinetics in Healthy and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-A001-002
Record Dates: First submitted 2012-08-21; First posted 2012-08-28 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: CNS
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Placebo comparator
- E2006 (Experimental)
  Interventions: Drug: E2006

INTERVENTIONS:
Drug: E2006 — Part A: 2.5 mg, 5 mg, 10 mg, 25 mg, 50 mg, and 75 mg E2006 administered as capsules
  Arms: E2006
Drug: Placebo comparator — E2006-matched placebo (Part A and Part B); Part B: dose level to be determined based on results of Part A, administered as capsules
  Arms: Placebo comparator

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, sequential, multiple-dose study. The study will be conducted in two parts: Part A (6 cohorts of healthy adults receiving evening dosing) and Part B (one cohort of elderly adults receiving evening dosing).

ELIGIBILITY:
Included:

* Healthy males or females, ages 18 to 55 years (Part A) or 65 to 80 years (Part B)
* Who report typical time in bed 7.5 to 9 hours
* Who report typical bedtime 22:00 - 24:00 and typical wake time 06:00 - 08:00
* Who report typical sleep latency of <= 30 minutes
* All females must be of non-childbearing potential, or subjects who have been sterilized surgically or who are otherwise proven sterile. Females must have a negative serum beta-human chorionic gonadotropin (Beta-hCG) test result at Screening and a negative urine pregnancy test at Baseline.
* Body mass index BMI > 18 and 32 kg/m2 at Screening

Excluded:

* Performed shift work within 2 weeks prior to Screening
* Had taken a flight across three or more time zones in the 7 days prior to Screening
* Female subjects who are nursing
* With a history of gastrointestinal surgery (hepatectomy, nephrectomy, digestive organ resection, etc.) that may affect PK profile of E2006
* With a known history of clinically significant drug or food allergies or presently experiencing significant seasonal allergy
* Hypersensitivity to the study drug or any of the excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events (AEs) | 28 days

SECONDARY OUTCOMES:
Plasma concentrations of E2006 | Part A up to 288 hours postdose; Part B: up to 324 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Dohwa Kim, Principal Investigator — Parexel
Locations (2):
- United States (2):
  - Parexel, California Clinical Trials, Culver City, California
  - Glendale, California